CLINICAL TRIAL: NCT00577902
Title: Nutritional Risk and Mucositis in Patients With Head and Neck Carcinoma Receiving Chemoradiation
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 41011
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Observation

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected and nutritional risk evaluated, using the Patient-Generated Subjective Global Assessment tool (PG-SGA). The PG-SGA and blood tests will be performed before, at the end of XRT treatment and four to six weeks after treatment is completed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: This is an observational study
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Head and neck cancer patients receiving chemoradiation

SUMMARY:
This study is being conducted to define the specific nutritional biomarkers and nutritional risk during the course of chemoradiation therapy for cancers of the head and neck. This prospective, longitudinal observational study is focused on specific antioxidants and B vitamins. The ORAC was selected as an index of overall antioxidant capacity. We chose to evaluate antioxidant status because administering antioxidants has been shown to reduce chemotherapeutic agent toxicities.

DETAILED DESCRIPTION:
The study will include 60, ≥18 year old patients (of both genders) with head and neck cancers receiving concurrent radiation and chemotherapy treatment. Patients with any pathologically proven head and neck squamous cell carcinoma, except those of the nasopharynx and sinus will be eligible, if there is no evidence of metastatic disease. Patients with previous chemotherapy or radiation treatment will be excluded. A Karnofsky performance status ≥60% or more is required. Patients with significant cardiac, chest or gastrointestinal comorbidities will be excluded, as will those who have had previous chemotherapy or radiation treatment. Patients may receive standard nutritional care, as needed.

This study will involve an examination of the patient to evaluate mucositis, collection blood samples for analysis of specific indicators of nutritional status and completion of questionnaire regarding food intake and functional status. Blood samples will be collected and brief questionnaires about diet and weight status will be completed at each of the three visits. Visits will occur before treatment begins, at the end of XRT treatment and 4-6 weeks after completion of XRT. Assessments for the presence and severity of mucositis and functional status (Karnofsky) will be done at each visit. All of the samples and data collection will be done at visits to clinic required for the patients' treatment. If it is necessary to obtain blood samples from the central venous catheter, this will be done using aseptic technique and will be performed by a nurse. In some instances, the information obtained as part of this project may be used to reduce side effects of therapy.

ELIGIBILITY:
Methodology. Patients presenting at the UAMS Head and Neck Clinic will be invited to participate in this study according to the inclusion criteria listed:

1. Age over 18 years,
2. Pathologically proven squamous cell carcinomas of the head and neck, except nasopharyngeal and sinus
3. Concurrent radiation and chemotherapy (taxotere/carboplatin)
4. Karnofsky score over60
5. Must receive radiation (IMRT)/chemotherapy at UAMS
6. No evidence of metastatic disease
7. No significant cardiac, chest, gastrointestinal or renal morbidities
8. No previous chemotherapy or radiation If they are considered eligible and agree to participate, the patients will be registered and sign informed consent form. Radiation and chemotherapy will commence on the same day. IMRT is the only modality of radiation allowed. Blood samples will be collected and nutritional risk evaluated, using the Patient-Generated Subjective Global Assessment tool (PG-SGA). The PG-SGA and blood tests will be performed before, at the end of XRT treatment and four to six weeks after treatment is completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the UAMS Head and Neck Clinic will be invited to participate in this study according to the inclusion criteria listed:
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2005-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To study baseline antioxidant capacity (ORAC), selected biomarkers of nutritional status and nutritional risk of patients beginning therapy for head and neck cancers.

SECONDARY OUTCOMES:
To assess antioxidant capacity, nutritional biomarkers and nutritional risk of patients during and after concurrent radiation and chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Hine, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States